CLINICAL TRIAL: NCT01293227
Title: The Effect of Intramedullary Locked Nail Versus Volar Locked Plating in the Treatment of Extra-articular and Minimally Displaced Intra-articular Distal Radius Fractures: A Prospective Randomized Trial.
Brief Title: WRx Distal Radius Wrist Fracture Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was withdrawn due to inadequete enrollment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Alexander Shin, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-005213
Record Dates: First submitted 2011-02-04; First posted 2011-02-10 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Wrist Fracture
Keywords: Wrist Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Surgical treatment of distal radius fractures — Surgical repair of distal radius fracture using either intramedullary locked nail or volar locked plate

SUMMARY:
This research project is a multi-year proposal, with the goals of answering and evaluating the following:

1. Does an intramedullary locking device applied in an extra-articular distal radius fracture improve post operative pain, diminish hospitalization, improve early return to activity and function compared to a volar locked plate?
2. Does an intramedullary locking device applied in an extra-articular distal radius fracture improve patient related outcome measures compared to a volar locked plate?

ELIGIBILITY:
Inclusion Criteria

The following criteria must be met to be enrolled:

1. Have a closed extra-articular distal radius fracture or a minimally displaced intra-articular component
2. Have a fracture classified as an AO Type A or C1 with or without an ulnar styloid fracture
3. Be a male or non-pregnant female at least 18 years of age.
4. Understand the requirements of the study and able to provide a written informed consent and comply with the study protocol
5. Have the ability to understand and provide written authorization for use and disclosure of personal health information
6. Have a fracture that can be closed reduced to acceptable radiographic parameters (minimum of neutral volar tilt, greater than or equal to 15 degrees of radial inclination and at least 10 mm of radial height as compared to the opposite side)

Exclusion Criteria

Subjects are excluded if:

1. Have any of the following conditions

   1. Concomitant contralateral or ipsilateral upper extremity fractures
   2. Ipsilateral ulna (excluding styloid) fracture
   3. Open, multifragmentary fracture
   4. Unstable distal radioulnar joint after fracture fixation
   5. Artery or Nerve injury secondary to fracture
2. Previous ipsilateral distal radius fracture in the 2 years prior to enrollment with deformity
3. Currently on chemotherapy or radiation therapy
4. History of a metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis
5. History of uncontrolled diabetes
6. History of active rheumatologic disease with deformity
7. History of chronic pain issues, psychiatric disorder which precludes reliable follow-up
8. Unable to provide consent for the study
9. Unable to make the follow-up appointments required of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain (to no pain) | Baseline to week 52 after surgery
  Postoperative pain will be monitored by recording of the consumption of narcotic pain medications converted to morphine equivalents. Participants will record medications taken in a Pain Diary. They will also be asked to complete a Visual Analog scale questionnaire regarding their pain.

SECONDARY OUTCOMES:
Change in range of motion measurements | Basline to week 52 after surgery
  Range of motion measurements will be measured using a goniometer and moving the hand and wrist into specific postitions.
Grip and Pinch | Baseline to week 52 after surgery
  Measurements of grip and pinch strength will be taken using a pinch gauge and a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States